CLINICAL TRIAL: NCT07367321
Title: Comparison of Onlay Mesh Repair and Sublay Mesh Repair in Umbilical Hernia Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Nurettin Şahin, Consultant General Surgeon, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSK-UMH-ONLAY-SUBLAY-2026
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Umbilical Hernia Repair; Onlay Mesh
Keywords: umbilical hernia repair; onlay mesh repair; sublay mesh repair

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either onlay mesh repair or sublay mesh repair in parallel groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Onlay Mesh Repair Group (Active Comparator): Patients undergoing elective umbilical hernia repair with onlay mesh placement on the anterior fascia.
  Interventions: Procedure: Onlay Mesh Repair
- Sublay Mesh Repair Group (Active Comparator): Patients undergoing elective umbilical hernia repair with sublay mesh placement beneath the fascia (retromuscular or preperitoneal plane).
  Interventions: Procedure: Sublay Mesh Repair

INTERVENTIONS:
Procedure: Onlay Mesh Repair — Umbilical hernia repair performed with mesh placement on the anterior fascia following primary fascial closure.
  Arms: Onlay Mesh Repair Group
Procedure: Sublay Mesh Repair — Umbilical hernia repair performed with mesh placement beneath the fascia in the retromuscular or preperitoneal plane.
  Arms: Sublay Mesh Repair Group

SUMMARY:
Umbilical hernia is a common condition that is frequently treated with surgical mesh repair to reduce recurrence rates. Among the commonly used techniques, onlay mesh repair and sublay mesh repair are widely performed; however, there is ongoing debate regarding their comparative effectiveness and safety.

The aim of this study is to compare onlay mesh repair and sublay mesh repair in patients undergoing elective umbilical hernia surgery, with respect to postoperative complications, recurrence rates, operative outcomes, and length of hospital stay. By evaluating clinical outcomes associated with each technique, this study seeks to contribute evidence to guide the selection of the most appropriate surgical approach for umbilical hernia repair.

DETAILED DESCRIPTION:
Umbilical hernia repair is one of the most commonly performed general surgical procedures. The use of prosthetic mesh has been shown to significantly reduce recurrence rates compared with primary suture repair. Among mesh-based techniques, onlay and sublay mesh repairs are frequently utilized, each with distinct technical characteristics and potential advantages and disadvantages.

In onlay mesh repair, the mesh is placed over the anterior fascia following primary fascial closure, whereas in sublay mesh repair, the mesh is positioned in the retromuscular or preperitoneal plane. While sublay mesh repair is often considered to provide better mesh integration and lower recurrence rates, it may be associated with longer operative times and increased technical complexity. Conversely, onlay mesh repair is technically simpler but has been associated with higher rates of wound-related complications in some studies. The optimal technique for umbilical hernia repair remains a subject of ongoing investigation.

This study is designed as a comparative clinical analysis of patients undergoing elective umbilical hernia surgery using either onlay mesh repair or sublay mesh repair. Adult patients who meet the eligibility criteria will be included. Demographic characteristics, hernia features, operative details, and perioperative outcomes will be recorded.

Primary outcome measures will include postoperative complication rates and hernia recurrence. Secondary outcome measures will include operative time, length of hospital stay, and early postoperative morbidity. Patients will be followed postoperatively according to standard clinical practice to assess surgical outcomes.

The results of this study are expected to provide comparative data on the safety and effectiveness of onlay and sublay mesh repair techniques in umbilical hernia surgery and to support evidence-based decision-making in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 90 years
* Patients diagnosed with small or medium-sized umbilical hernia according to the European Hernia Society (EHS) classification
* Patients scheduled for elective umbilical hernia surgery
* Patients who provide written informed consent

Exclusion Criteria:

* Patients younger than 18 years or older than 90 years
* Patients undergoing emergency umbilical hernia surgery
* Patients with bowel obstruction
* Patients with chronic kidney failure
* Patients with a history of previous abdominal surgery involving the stomach, duodenum, small intestine, or colon

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complication Rate | Within 30 days after surgery
  Postoperative complications occurring after umbilical hernia surgery, including surgical site infection, seroma, hematoma, wound-related complications, and other procedure-related adverse events.

SECONDARY OUTCOMES:
Hernia Recurrence Rate | Up to 6 months after surgery
  Occurrence of recurrent umbilical hernia detected during postoperative follow-up.
Postoperative Pain Score | First 7 days after surgery
  Postoperative pain assessed using the Visual Analog Scale for Pain, ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores indicate worse pain severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No